CLINICAL TRIAL: NCT03734770
Title: Patient's Preferences About Subcutaneous or Vaginal Progesterone Administration for Luteal Phase Support: Prospective Randomized Trial.
Brief Title: Patient's Preferences About Subcutaneous or Vaginal Progesterone Administration for Luteal Phase Support
Acronym: PROPER-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Simone Garzon, Principal Investigator, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROPER-1
Record Dates: First submitted 2018-10-31; First posted 2018-11-08 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Progesterone; Luteal Phase Support; In Vitro Fertilization
Keywords: progesterone; subcutaneous; vaginal; luteal phase support; in vitro fertilization

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous progesterone (Active Comparator): After standard stimulating protocol for IVF, beginning on the day of oocyte retrieval allocated patients receive subcutaneous progesterone (Pleyris, IBSA Farmaceutici, Italia) 25 mg one time per day (every day at the same time, according to patient's availability and preference) for at least 8 gestational weeks or confirmation of a negative pregnancy test performed 14 days after oocyte retrieval.
  Interventions: Drug: Subcutaneous Progesterone
- Vaginal progesterone (Active Comparator): After standard stimulating protocol for IVF, beginning on the day of oocyte retrieval allocated patients receive micronized vaginal progesterone (Progeffik, EFFIK Spa, Italia) 200 mg three times per day (every 8 hours) for at least 8 gestational weeks or confirmation of a negative pregnancy test performed 14 days after oocyte retrieval.
  Interventions: Drug: Vaginal progesterone

INTERVENTIONS:
Drug: Subcutaneous Progesterone — Subcutaneous progesterone (Pleyris, IBSA Farmaceutici, Italia) 25 mg one time per day (every day at the same time, according to patient's availability and preference).
  Arms: Subcutaneous progesterone
Drug: Vaginal progesterone — Micronized vaginal progesterone (Progeffik, EFFIK Spa, Italia) 200 mg three times per day (every 8 hours).
  Arms: Vaginal progesterone

SUMMARY:
Luteal phase support in "in vitro fertilization" (IVF) cycles has been shown to improve pregnancy rates and became a standard of treatment, and progesterone is the first choice considering its safety profile and effectiveness. There are many studies demonstrating that vaginal progesterone is equally efficacious and better tolerated compared to intramuscular progesterone for luteal phase support in IVF cycles. Conversely, although different studies showed that subcutaneous progesterone is equally efficacious compared to vaginal progesterone, patient use satisfaction and compliance were less studied with few evidences are available, that may guide the choice of vaginal progesterone instead of subcutaneous progesterone and other way around. Considering the paucity of published data about the patient's preference and use satisfaction about subcutaneous progesterone, the investigators will conduct a prospective randomized study aimed to compared adverse effects rates, impact on quality of life, use satisfaction and administration preference in women undergoing luteal phase support with vaginal progesterone versus subcutaneous progesterone during IVF cycles, that may guide the choice for luteal phase support in IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women candidate to undergo fresh IVF cycles

Exclusion Criteria:

* day-3 follicle-stimulating hormone (FSH) levels over 15 IU/L
* clinically relevant systemic disease (e.g., uncontrolled thyroid and adrenal dysfunction, an organic intracranial lesion such as a pituitary tumor, insulin-dependent diabetes mellitus, cancers)
* hypersensitivity to any of the study drugs
* contraindications to use the study drugs
* surgical or medical condition that would interfere with absorption, distribution, metabolism, or excretion of the study drugs

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Grade of use satisfaction reported by the patients | At the human chorionic gonadotropin test performed after 14 days of progesterone use
  Patients will be asked how satisfied they are by the use of progesterone product that they receive in the luteal phase. Their satisfaction responses will be recorded on a scale of 1 to 3, with 1 being ''least satisfied'' and 3 being ''most satisfied'.
Grade of quality of life impairment reported by the patients | At the human chorionic gonadotropin test performed after 14 days of progesterone use
  Patients will be asked whether work life, social life, sexual life, and personal hygiene are perceived impaired by the progesterone treatment that they received. The answer for each item is "yes" or "no".
Adverse effects (AEs) | At the human chorionic gonadotropin test performed after 14 days of progesterone use
  Patients will be asked to report experienced AEs. The investigated AEs are sleepiness, dizziness, headache, bowel dysfunctions, breast pain/tension, weight changes, mood disorders, skin irritation, and vaginal discharge.
  The answer for each item is "yes" or "no".

SECONDARY OUTCOMES:
Progesterone administration route that the patients prefer | At the human chorionic gonadotropin test performed after 14 days of progesterone use
  Patients of subcutaneous progesterone arm and who had previously used vaginal progesterone will be asked which administration route they prefer.
Implantation rate | At the human chorionic gonadotropin test performed after 14 days of progesterone use
  Rate of positive human chorionic gonadotropin test
Clinically pregnancy rate | At 6 week from oocyte retrieval
  Rate of evolving pregnancy at ultrasound
live birth rate | At nine months from oocyte retrieval
  Rate of baby delivered after 24 gestational weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simone Garzon, M.D., Principal Investigator — Universita di Verona; Rossana Di Paola, M.D., Principal Investigator — Universita di Verona; Antonio Simone Laganà, Principal Investigator — Università degli Studi dell'Insubria; Francesca Parissone, M.D., Principal Investigator — Universita di Verona; Stefano Zaffagnini, M.D., Study Director — AOUI Verona; Massimo Franchi, M.D., Study Director — Universita di Verona; Ricciarda Raffaelli, M.D., Principal Investigator — Universita di Verona
Locations (1):
- AOUI Verona - University of Verona - Department of Obstetrics and Gynecology, Verona, Italy

IPD SHARING:
Plan to Share IPD: No